CLINICAL TRIAL: NCT02351492
Title: Diagnostic Pathway for Surgical Patients With Suspected Bile Duct Obstruction
Brief Title: Radiological Investigation of Bile Duct Obstruction
Acronym: RIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 221/13
Record Dates: First submitted 2015-01-07; First posted 2015-01-30 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Gallstone Disease
Keywords: Bile duct obstruction; intraoperative cholangiography; MRCP
MeSH Terms: conditions — Cholelithiasis; Cholestasis | interventions — Cholecystectomy; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecystectomy and intraoperative cholangiography (Active Comparator): Patients with suspected bile duct obstruction intraoperative cholangiography (IOC) to investigate bile ducts.
  Interventions: Procedure: Cholecystectomy and intraoperative cholangiography; Device: catheter
- Magnet resonance cholangio-pancreaticography (Active Comparator): Patients get Magnet resonance cholangio-pancreaticography (MRCP) first. In case of detected gallstones, removal of the stones by endoscopic retrograde cholangiopancreaticography will be performed before gallbladder removal.
  Interventions: Procedure: Magnet resonance cholangio-pancreaticography; Device: magnet resonance imaging

INTERVENTIONS:
Procedure: Cholecystectomy and intraoperative cholangiography — Patients with suspected bile duct obstruction intraoperative cholangiography IOC to investigate bile ducts.
  Other Names: IOC
  Arms: Cholecystectomy and intraoperative cholangiography
Procedure: Magnet resonance cholangio-pancreaticography — Patients get Magnet resonance cholangio-pancreaticography MRCP first. In case of detected gallstones, removal of the stones by endoscopic retrograde cholangiopancreaticography will be performed before gallbladder removal.
  Other Names: MRCP
  Arms: Magnet resonance cholangio-pancreaticography
Device: magnet resonance imaging — Patients get Magnet resonance cholangio-pancreaticography MRCP first. In case of detected gallstones, removal of the stones by endoscopic retrograde cholangiopancreaticography will be performed before gallbladder removal.
  Other Names: MRI
  Arms: Magnet resonance cholangio-pancreaticography
Device: catheter — Patients with suspected bile duct obstruction intraoperative cholangiography IOC to investigate bile ducts.
  Arms: Cholecystectomy and intraoperative cholangiography

SUMMARY:
Patients with gallstone disease should be checked whether a common bile duct (CBD) stone could be present. In case of a certain suspicion for CBD stones further investigations should be performed. This can either be done by magnetic resonance cholangio-pancreaticography (MRCP) or by intraoperative cholangiography. The study investigates which pathway would be favorable in regard of an early hospital demission.

DETAILED DESCRIPTION:
Patients with gallstone disease and suspected bile duct obstruction can be investigated either with a magnetic resonance cholangio-pancreaticography (MRCP) prior to gallbladder removal or with an intraoperative cholangiography during cholecystectomy. When detecting an common bile duct (CBD) stone in MRCP, normally endoscopic removal is performed before an operation. When the CBD stone is detected during gallbladder removal instead, endoscopic retrograde cannulation of the pancreatic duct (ERCP) will follow after the operation. Investigators hypothesize that direct operation shortens the length of hospital stay. Therefore investigators randomize patients with elevated Bilirubin, elevated liver enzymes (two of the following: aspartate transaminase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyltransferase (gGT) or AP), suspected CBD stones in ultrasound or dilated common bile ducts either in MRCP first or operation first pathway. All data (patient admission to discharge, ...) will be entered in an online database

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting as regular admission or at the emergency department (ED) with cholecystolithiasis and suspected CBD stones. The indication for CBD investigation requires one of the following features:

  i. Elevated bilirubin ii. ASAT/ALAT or gGT or aP above the normal range (two of them) iii. Choledocholithiasis in ultrasound iv. Dilated bile ducts in ultrasound
* Written informed consent

Exclusion Criteria:

* Age under 18 years
* Patients with biliary pancreatitis (due to the fact that conservative treatment is initiated before gallbladder removal and therefore leads to a prolonged hospital stay)
* Septic patients due to cholangitis
* Patients unable to consent
* Patients with medical conditions preventing surgery
* Pregnancy
* Radiologically proven CBD stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-05; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Length of Hospital stay | number of days patient spent in hospital assessed at discharge day, on average 8 days
  Time of hospital entry to time of patient dischargeable, according to stuff surgeon. Dates will be entered in an online database, which is also used for randomisation.

SECONDARY OUTCOMES:
Costs of Hospital stay | days in hospital assessed at hospital discharge day, on average 8 days
  Computed by the financial departments of each involved hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christian A. Nebiker, MD, PD Dr., Principal Investigator — Kantonsspital Aarau
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Staubli SM, Kettelhack C, Oertli D, von Holzen U, Zingg U, Mattiello D, Rosenberg R, Mechera R, Rosenblum I, Pfefferkorn U, Kollmar O, Nebiker CA. Efficacy of intraoperative cholangiography versus preoperative magnetic resonance cholangiography in patients with intermediate risk for common bile duct stones. HPB (Oxford). 2022 Nov;24(11):1898-1906. doi: 10.1016/j.hpb.2022.05.1346. Epub 2022 Jun 18. PMID 35817694